CLINICAL TRIAL: NCT06841328
Title: Fertility Enhancement Through Regenerative Treatment in Ovaries and Testes: (FERTILE): Prospective Observational Study Evaluating Safety and Efficacy
Brief Title: Fertility Enhancement Through Regenerative Treatment in Ovaries and Testes
Acronym: FERTILE
Status: Recruiting | Type: Observational
Sponsor: Jumeirah American Clinic (Other)
Responsible Party: Principal Investigator, Ranjith Ramasamy, Consultant Urologist, Jumeirah American Clinic
Other Study IDs: 002
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Gonadal Dysfunction; Gonadal Failure; Azoospermia; Testosterone Deficiency; Stem Cells; Hypogonadism, Male
Keywords: Premature Ovarian Failure; Testicular Failure; low testosterone; Stem cell therapy; Exosomes
MeSH Terms: conditions — Gonadal Disorders; Azoospermia; Eunuchism; Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Male: Male patients aged 20 to 50 years. Diagnosed with testicular failure (low testosterone) or hypogonadism (impaired gonadal function), or azoospermia due to production defect (no sperm in ejaculate)
  Interventions: Procedure: Stem cells
- Female: Female patients aged 20 to 50 years. Diagnosed with premature ovarian failure (POF) or ovarian insufficiency, confirmed through clinical, hormonal, and imaging assessments.
  Interventions: Procedure: Stem cells

INTERVENTIONS:
Procedure: Stem cells — The administration of stem cell or stem cell-derived exosome therapy as a regenerative treatment for gonadal failure in both men and women. The intervention involves a single intra-gonadal injection (testicular or ovarian) of adipose-derived stem cells (ADSCs) or exosomes.

SUMMARY:
This study investigates the safety and efficacy of stem cell or stem cell-derived exosome therapy for gonadal failure, including testicular failure, hypogonadism, ovarian insufficiency, and premature ovarian failure (POF). Conducted at First IVF Clinic, Dubai, it will include 60 participants (30 males, 30 females) aged 20-50 years who have not responded to conventional treatments such as HRT, TRT, or ART.

Participants will receive intra-gonadal (testicular or ovarian) injections of stem cells or exosomes, with follow-ups at 3, 6, 9, and 12 months to monitor hormonal changes, gonadal function, and potential adverse effects. The study aims to determine whether regenerative therapy can restore hormone production, enhance reproductive function, and regenerate gonadal tissue, providing a novel, culturally appropriate fertility treatment in the UAE, where donor sperm and eggs are not permitted.

By bridging the gap between preclinical research and clinical application, this study could offer new hope to individuals with gonadal failure, advancing the field of regenerative reproductive medicine.

DETAILED DESCRIPTION:
Background and Rationale:

Testicular and ovarian failure, often called 'gonadal failure,' occurs when the testes or ovaries lose their ability to produce gametes. Both lead to reduced fertility and hormonal deficiencies, significantly impacting an individual's health and quality of life. Conventional treatments such as hormone replacement therapy (HRT) help alleviate symptoms but do not restore fertility.

Surgical options (testicular sperm retrieval, ultrasound-guided egg retrieval) are found to be helpful for some. However, they are not uniformly successful 11. Surgeries (testicular biopsies) always carry risks such as risk of bleeding or infection and lack of guaranteed success 12. Clinicians are exploring less invasive alternatives like stem cell-based therapies, including adipose-derived stem cells (ADSCs) and exosomes. Stem cells or stem cell-derived exosome therapy offers a promising regenerative approach for restoring gonadal function by enhancing tissue repair, stimulating folliculogenesis or spermatogenesis, modulating hormonal balance, and improving overall reproductive potential in individuals with testicular or ovarian failure.

This study assesses the safety and efficacy of intra-gonadal (testicular or ovarian) stem cells or stem cell-derived exosome injection for patients with testicular and ovarian failure who have not responded to conventional treatments. ADSC therapy has been studied in humans for related conditions like ovarian insufficiency and POF (Premature ovarian failure)6. It has shown encouraging results in repairing damaged tissues and improving hormonal function, showing early successes that provide hope for its potential. This research assumes even greater importance in the UAE, where donor sperm and eggs are not permitted due to religious and legal restrictions 13. Testing the safety and long-term efficacy of ADSC therapy for gonadal failure in the UAE could provide a groundbreaking, culturally appropriate solution for individuals facing reproductive challenges, giving them new opportunities for treatment and a renewed sense of hope.

The Bioscience Institute, a DHA-approved facility, will provide the stem cells or stem cell-derived exosomes under an existing Memorandum of Understanding (MOU) with the First IVF Clinic and Day Surgery Center. The stem cells or stem cell-derived exosomes will be extracted and produced in an off-site laboratory (Bioscience Institute) and undergo sterility, cell count, and viability check before being prepared for administration back into the patient. The manufacturing process follows CGTP. The cells will be injected directly into the testes and ovaries under anesthesia.

Study Objectives

* Primary Objective:

  1. To evaluate the safety and efficacy of intraovarian or intratesticular injections of stem cells or stem cell-derived exosomes in restoring gonadal function, as measured by hormonal changes (testosterone, estradiol, FSH, AMH) and reproductive capacity from baseline to post-treatment.
* Secondary Objectives:

  1. Assess gonadal tissue regeneration using imaging techniques.
  2. Monitor long-term treatment effects at follow-up points
  3. Document any adverse events or complications related to stem cell or exosome therapy, such as fibrosis, infection, or immune reactions.
  4. Evaluate functional outcomes such as spermatogenesis in men (via semen analysis) and ovarian follicular activity in women (via antral follicle count and menstrual cycle regularity).
  5. Compare the effects of stem cells vs. stem cell-derived exosomes in improving gonadal function and hormone levels.

Study Design and Objectives This open-label, single-arm, pilot observational study will serve as a preliminary investigation into the use of adipose-derived stem cells (ADSCs) or stem cell-derived exosomes for treating gonadal failure in both men and women. The study's primary focus will be on assessing safety and feasibility, while also gathering initial efficacy data to support future large-scale trials.

Study Population The study will enroll 60 adults (30 males, 30 females) aged 20 to 50 years diagnosed with gonadal failure, including testicular failure, hypogonadism, ovarian insufficiency, or premature ovarian failure (POF). Participants must have failed or experienced suboptimal responses to conventional treatments, such as hormone replacement therapy (HRT), testosterone replacement therapy (TRT), or assisted reproductive technologies (ART).

Recruitment will take place at First IVF Clinic, Dubai, where participants are actively receiving evaluation and treatment for gonadal failure. The inclusion and exclusion criteria will ensure that the study targets individuals most likely to benefit from therapy while prioritizing patient safety.

Sample Size Rationale A sample size of 60 participants was selected based on the exploratory nature of the study. The primary objective is to assess the feasibility, safety, and preliminary efficacy of stem cell or exosome therapy while providing sufficient data to inform the design of future, larger trials. Given the clinic's patient population, recruiting 60 participants over the planned two-year study period is considered achievable.

Study Procedures

1. Informed Consent Participants will receive detailed information about the study, including its risks and potential benefits, and will provide written consent prior to enrollment.
2. Baseline Assessments

   Before treatment, participants will undergo comprehensive baseline testing, including:

   Hormonal blood tests (Testosterone, Estradiol, FSH, AMH)

   Ultrasound imaging (AFC for ovaries, testicular volume for testes)

   Semen analysis (for male participants, if applicable)

   Medical history review and general health evaluation
3. Therapeutic Administration

   For ADSCs:

   ADSCs will be harvested via minimally invasive liposuction from the participant's own adipose tissue.

   The cells will be processed, purified, and prepared for injection into the ovaries (females) or testes (males).

   For Exosomes:

   Exosomes will be derived from stem cells, isolated, and purified before administration.

   The injections will follow the same procedure as stem cell therapy, ensuring targeted delivery into the gonads.

   Injection Procedure:

   Ovarian injections: Administered via direct intraovarian injection. Testicular injections: Administered via direct intratesticular injection in rete testis.
4. Follow-Up Monitoring

Participants will be monitored immediately post-injection for any adverse reactions and will return for regular follow-ups at 3, 6, 9, and 12 months to assess:

Data Collection and Analysis Collected data will be analyzed to evaluate primary and secondary outcomes.

Primary Outcome:

Hormonal level changes from baseline to 12 months post-treatment.

Secondary Outcomes:

Changes in gonadal tissue structure (AFC, testicular volume). Functional improvements (spermatogenesis, menstrual cycle regulation). Incidence of adverse events (infection, fibrosis, immune response). Surgical sperm retrieval and Egg retrieval success

Ethical Considerations This study will adhere to strict ethical standards for clinical research.

Ethics Committee Review: The protocol will be reviewed and approved by an independent ethics board.

Informed Consent: Participants will have full autonomy to decide on participation and may withdraw at any time without affecting their standard medical care.

Confidentiality: All patient data will be anonymized and stored securely to ensure privacy.

Expected Outcomes

This study aims to provide early evidence on the safety and potential efficacy of stem cell or exosome therapy for gonadal failure. If successful, participants are expected to show:

Improvements in hormone levels and reproductive function. Gonadal tissue regeneration, restoring follicular activity or spermatogenesis. Minimal adverse effects, confirming safety and feasibility. The findings from this study will help guide future, larger-scale trials and contribute to the development of regenerative therapies for gonadal failure, offering a novel and culturally appropriate solution for fertility preservation in the UAE.

ELIGIBILITY:
Male patients:

* Male patients aged 20 to 50 years.
* Diagnosed with testicular failure (low testosterone) or hypogonadism (impaired gonadal function), or azoospermia (no sperm in ejaculate)
* Suboptimal response to conventional treatments, such as testosterone replacement therapy (TRT) or fertility-enhancing medications (Clomiphene citrate or anastrozole).
* General good health without significant contraindications to stem cell or stem cell-derived exosome therapy.
* Willing and able to provide informed consent and comply with the study protocol.
* Patients who have been evaluated for testicular failure and are seeking further treatment.

Female patients:

* Female patients aged 20 to 50 years.
* Diagnosed with premature ovarian failure (POF) or ovarian insufficiency, confirmed through clinical, hormonal, and imaging assessments.
* Failure or suboptimal response to conventional treatments, such as hormone therapy.
* General good health without significant contraindications to stem cell or stem cell-derived exosome therapy.
* Willing and able to provide informed consent and comply with the study protocol.
* Patients who have been evaluated for ovarian failure are seeking further treatment.

Exclusion criteria

* Severe comorbid conditions, such as advanced cardiovascular disease, renal failure, or uncontrolled diabetes.
* Active malignancies or history of cancer within the past 5 years.
* Active infections or systemic inflammatory conditions.
* History of testicular surgery or trauma that could interfere with the study outcomes.
* Use of anticoagulants or medications that may contraindicate stem cell or stem cell-derived exosome therapy.
* Participation in another investigational drug or treatment study within the past 6 months.
* Contraindications to stem cell or stem cell-derived exosome therapy, such as immune deficiencies or allergies to any treatment components.
* Severe neurological disorders or cognitive impairment may limit the ability to provide informed consent or follow study instructions.
* Any condition that, in the investigator's opinion, could interfere with the study or pose an undue risk to the patient.
* Women with a primary diagnosis of psychogenic ovarian dysfunction or infertility.
* History of ovarian surgery or trauma that could interfere with the study outcomes.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of adult male and female patients aged 20 to 50 years who are diagnosed with testicular or ovarian failure and are seeking treatment at First IVF and Day Surgery Center. Participants will be recruited from the pool of patients under the care of the PI or the co-Is. Eligibility will include individuals with confirmed testicular or ovarian failure based on clinical, hormonal, and imaging criteria who have not responded adequately to conventional treatments such as hormone therapy (HT).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in reproductive capacity | 12 months
  We will evaluate hormonal changes (testosterone, estradiol, FSH, AMH) and sperm parameters

SECONDARY OUTCOMES:
Gonadal Function | 12 months
  Evaluate functional outcomes such as surgical sperm retrieval success and ovarian follicular activity in women (via antral follicle count and egg retrieval success)

OTHER OUTCOMES:
Adverse Effects | 12 months
  Document any adverse events or complications related to stem cell or exosome therapy, such as fibrosis, infection, or immune reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Ranjith Ramasamy, MD, Principal Investigator — Jumeirah American Clinic
Locations (1):
- First IVF and Day Surgery Center, Dubai, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
The study will involve the collection of individual participant data (IPD) related to adult male and female patients aged 20 to 50 years diagnosed with testicular or ovarian failure who are seeking treatment at First IVF and Day Surgery Center. The specific IPD that will be shared includes:
  1. De-identified Data to be Shared Demographic Data: Age, sex, and relevant medical history (without personal identifiers).
     Clinical Data: Diagnosis of testicular or ovarian failure, including clinical presentation and duration of symptoms.
     Hormonal and Imaging Data: Laboratory test results (e.g., hormone levels such as FSH, LH, testosterone, estrogen) and imaging findings confirming the diagnosis.
     Treatment and Response Data: Information on previous hormone therapy (HT) and response status.
     Outcome Measures: Treatment efficacy, adverse events, and follow-up assessments.
  2. Data Not to be Shared Personal identifiers such as names, contact details, and specific identifying information.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: May 2026 to May 2028
Access Criteria: Upon formal request to PI

REFERENCES:
- [Background] Zafardoust S, Kazemnejad S, Darzi M, Fathi-Kazerooni M, Rastegari H, Mohammadzadeh A. Improvement of Pregnancy Rate and Live Birth Rate in Poor Ovarian Responders by Intraovarian Administration of Autologous Menstrual Blood Derived- Mesenchymal Stromal Cells: Phase I/II Clinical Trial. Stem Cell Rev Rep. 2020 Aug;16(4):755-763. doi: 10.1007/s12015-020-09969-6. PMID 32198596